CLINICAL TRIAL: NCT01480518
Title: Analysis of GGAA-Microsatellites in Ewing Sarcoma
Brief Title: Biomarkers in Tissue Samples From Patients With Ewing Sarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEWS11B2; COG-AEWS11B2 (Other: Children's Oncology Group); AEWS11B2 (Other: Children's Oncology Group); NCI-2012-00083 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Sarcoma
Keywords: localized Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Comparative Genomic Hybridization; Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: comparative genomic hybridization
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphic microsatellite marker analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with Ewing sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To describe the spectrum of GGAA-microsatellite polymorphisms at specific loci in genomic DNA prepared from Ewing sarcoma tumor specimens.
* To determine if there are differences in GGAA-microsatellite polymorphisms in genomic DNA prepared from Ewing sarcoma tumor specimens as compared to non-afflicted European and African normal genomic DNA.
* To determine if GGAA-microsatellite polymorphisms at specific loci in genomic DNA prepared from Ewing's sarcoma tumor specimens correlates with disease outcome in patients treated on COG protocol AEWS0031.
* To determine whether whole-genome amplification introduces alterations in GGAA-microsatellites as compared to non-amplified genomic DNA.

OUTLINE: Genomic PCR is used to amplify the microsatellites in the NR0B1 and GSTM4 promoters. In addition to determining microsatellite size, each microsatellite is sequenced following cloning into the pCR4 vector (Invitrogen) using standard topoisomerase cloning protocols.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Specimens from patients with Ewing sarcoma used for protocol COG-AEWS08B1

  * Obtained from patient samples taken from patients enrolled on COG-AEWS0031
  * Whole genome-amplified DNA will be used

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ewing sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lessnick, MD, PhD, Principal Investigator — University of Utah